CLINICAL TRIAL: NCT05808413
Title: Promoting Protection of Others to Increase Future COVID-19 Booster Shot Vaccination Intentions in Younger Adult Canadians: Evaluating the Efficacy of Short Video-based Interventions
Brief Title: Exploring the Effect of Video Interventions on Intentions for Continued COVID-19 Vaccination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Zeev Rosberger, Senior Investigator, Sir Mortimer B. Davis - Jewish General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2023-3198
Record Dates: First submitted 2023-04-07; First posted 2023-04-11 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Vaccine Refusal; COVID-19
Keywords: Vaccine Hesitancy; Vaccine Decision Making
MeSH Terms: conditions — Vaccination Refusal; COVID-19; Vaccination Hesitancy

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of: 1) a control video, 2) the control + an altruistic video, or 3) the control + altruistic video + individualistic video. A 1:1:1 randomization ratio will be used.
Who Masked: Investigator
Masking Description: The survey company, Dynata, will collect all data and manage group assignments. Participants' intervention group assignments will be unavailable to the investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Informational Video (Active Comparator): Participants will watch a 1-minute video detailing the impact vaccination has had on the COVID-19 pandemic, where accurate information on vaccination can be found, and the convenience of vaccination.
  Interventions: Behavioral: Informational Video
- Informational + Altruistic Video (Experimental): Participants will first watch the 1-minute informational video before watching an additional 40-second video eliciting altruistic motivations for vaccination. The purpose of this arm is to test whether altruistic messages are efficacious to increase vaccine intentions beyond providing only vaccine information.
  Interventions: Behavioral: Informational Video; Behavioral: Altruistic Video
- Informational + Altruistic + Individualistic Video (Experimental): Participants will watch the 1-minute informational video, the 40-second altruistic video, and an additional 40-second video eliciting individualistic motivations for vaccination. This arm will be used to test if combined altruistic and individualistic messages provide a greater effect than providing only vaccine information.
  Interventions: Behavioral: Informational Video; Behavioral: Altruistic Video; Behavioral: Individualistic Video

INTERVENTIONS:
Behavioral: Informational Video — This video emphasizes that vaccination against COVID-19 continues to be important, highlights the importance of seeking accurate information, and provides statistics about the estimated number of lives saved by vaccination and reported adverse events following vaccination in Canada.
Behavioral: Altruistic Video — This video presents a vignette about a young adult woman who has many social interactions during her daily life. It shows that her decision to stay up-to-date on COVID-19 vaccination could help to protect those people she comes into contact with, who may be at greater risk from COVID-19 infection. Statistics are used to show that up to one-in-four people in Canada have underlying conditions that make them more vulnerable to COVID-19, and to quantify the number of surgeries that were delayed by pandemic-related disruptions.
  Arms: Informational + Altruistic + Individualistic Video; Informational + Altruistic Video
Behavioral: Individualistic Video — This video presents a vignette about a young adult man who is very health-conscious. He is unsure about staying up-to-date on COVID-19 vaccination until he learns that COVID-19 infection can have serious and disruptive consequences even if someone is younger. Statistics are used to quantify the increased risk of severe symptoms in young adults who are not up-to-date on vaccination.
  Arms: Informational + Altruistic + Individualistic Video

SUMMARY:
While COVID-19 vaccine uptake has generally been high in Canada, with 83.4% of the total population having received the first two doses (i.e., primary series), additional "booster" uptake has been slower, especially among young adults aged 18-39. Throughout the pandemic, young adults have experienced less personal risk from COVID-19 infection and this has led to lower motivation to vaccinate when it is recommended. Achieving high rates of up-to-date vaccine coverage is important in this group to anticipate new variants and waves of infection and changes to recommendations which might include annual or seasonal vaccination. Three video interventions, intended to motivate Canadian young adults to adopt positive intentions toward continued COVID-19 vaccination, will be developed and tested: an informational comparison video, an altruistic video, and an individualistic video. Participants will be 3300 Canadian younger adults who will be randomly assigned to watch these videos. The first arm will only receive the informational video, the second arm the informational and altruistic videos, and the third arm the informational, altruistic, and individualistic videos. All participants will complete a brief online survey before and after viewing the assigned video(s). The goal of the study is to examine the efficacy of altruistic and individualistic messages, beyond informational messages, in increasing intentions for COVID-19 vaccination in this age group.

DETAILED DESCRIPTION:
The COVID-19 vaccine has significantly reduced mortality from the COVID-19 disease, and relieved the pressure on society, the economy, and the healthcare system caused by the pandemic. However, waning immunity and the emergence of new, vaccine-evasive variants like Omicron have necessitated additional vaccine doses, or "booster shots". Similar to trends for COVID-19 vaccination and other routine vaccinations, young adults (aged 18-39) have demonstrated lower uptake of booster vaccination, and evidence suggests that public health recommendations are no longer translating to vaccine uptake. This study will examine the efficacy of altruistic and individualistic messages over informational messages in increasing vaccine intentions in this age group.

This study has four primary objectives:

1. Estimate pre- to post-intervention changes in COVID-19 vaccine intentions of a altruistic video intervention.
2. Estimate pre- to post-intervention changes in COVID-19 vaccine intentions of a combined altruistic + individualistic video
3. Estimate between-group (altruistic vs. vaccine-informational) differences in COVID-19 vaccine intentions post-intervention
4. Estimate the between-group (altruistic + individualism vs. vaccine-informational) differences in COVID-19 vaccine intentions post-intervention

In addition, there is an exploratory, multivariable objective:

1. To estimate the multivariable associations of vaccine intentions in each intervention group.

A survey will be administered online to a sample of Canadian residents, aged 18-39, in both English and French. Participants will be drawn from a database panel provided by Dynata, a multinational first-party data and insight platform. Dynata's use of Canadian census data from Statistics Canada and quota-based sampling will ensure that the sample will closely match the Canadian population in terms of age (18-29, 30-39), sex, first language English/French, population density (i.e., urban vs. rural), and household income. Dynata will send invitations in various forms (e.g., e-mail invitations, text messages and in-app alerts) to recruit eligible participants from their existing panel (individuals who have signed with Dynata and have expressed willingness to receive invitations to various appropriate surveys) until recruitment goals and quotas are met.

To calculate the required sample size for the within-participant change in vaccine hesitancy (i.e., pre-post intervention) hesitancy towards continuing to receive booster vaccination was estimated at about 70% in the sample population. This estimate of the hesitancy rate at time of writing was based on seasonal influenza vaccination uptake in the target age range (between 20-25%) and uptake of COVID-19 booster vaccination in the past 6 months (9.2 - 14.5%) accounting for a gradual increase in uptake observed over time. Informed by results of a previous two-arm RCT conducted by this research team (NCT04960228) that included a video-based intervention and an active control group, it is estimated that the intentions in the control group will increase from 30% to 33% and in the intervention groups from 30% to 39%. To detect a 6% difference in intentions between arms, at a 95% confidence level (for a two-sided significance level α=0.025) and a desired statistical power of 80%, it was calculated that the minimum required number of participants per arm would be N=1005. 1:1:1 randomization will be used the three between groups. Thus, one-third of the participants will be allocated to each intervention group. Including 95 additional participants per arm to account for possible inattentive responders, the total sample required for this study is 3300 participants i.e., 1100 in each of the two experimental groups and 1100 in the active comparator group.

Stratified randomization will be used for first language (English/French), sex (male/female), population density (Urban/rural) and household income (<$75,000 / >$75,000) to allocate participants to either intervention arm. Within each stratum, a random concept picker approach will be used to ensure a 1:1:1 allocation using groups of three participants. Correspondingly, the first participant of a group will be randomly allocated to one of the three study arms, the second randomly assigned to one of the two remaining arms, and the third to the remaining arm. If a participant does not finish the survey (incomplete data), that place in the group will be allocated to the next participant. Thus, the quota in each stratum will be filled in groups of three and ensure a balanced group allocation throughout data collection.

The initial online survey will be approximately 12 minutes in length and will be available in both French and English. After reading the introductory statement of the study, participants will be asked for their consent to take part in the survey. Those who consent to participate will be invited to go to the next page and start completing the survey. Participants will first be asked to answer several socio-demographic questions and will be asked to choose their current Precaution Adoption Process Model stage for continued COVID-19 vaccination. Participants will then watch the assigned intervention. After viewing this content, to ensure that participants paid attention, participants will answer questions about the interventions to check their attention. Finally, participants will: 1) once again be asked to choose their vaccine decision-making stage; 2) be asked questions regarding previous vaccination history (e.g., seasonal influenza, COVID-19), lifestyle factors, self-perceived health status, personal history of SARS-CoV-2 infection, and preferred health-information channels; and 3) complete validated scales regarding, empathy, distress, intolerance of uncertainty, individualism and collectivism, COVID-19 pandemic fatigue, intellectual humility, and social desirability.

To test within-participant outcomes (Objectives 1 and 2), McNemar's test will be used to compare paired (pre and post-intervention) proportions. Additionally, exact tests of symmetry comprising of multiple pairwise McNemar tests to estimate pre-post changes in vaccine intentions. Adjusted p values for multiple comparisons, odds ratios (OR) and Cohen's g effect sizes will be reported. For each study group, the significant transitions between vaccine intention stage pairs will be used for calculating the total number of participants that changed towards increased vaccination intentions (e.g., from undecided to decided to). To test between-group outcomes (Objectives 3 and 4), the Chi-square test will be used to examine differences in PAPM stage proportions between intervention groups.

For the exploratory objective, Structural Equation Modelling will be used to identify multivariable associations of vaccine intentions (e.g., collectivism, empathy, intolerance of uncertainty) and to control for the potential effect of other factors (e.g., sociodemographics, psychosocial factors, previous influenza vaccination, lifestyle factors).

ELIGIBILITY:
Inclusion Criteria:

* Residing within Canada
* Aged between 18 and 39.

Exclusion Criteria:

-

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3567 (Actual)
Dates: Start 2023-06-06 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Vaccine Intentions | Pre- and post-intervention, within the same survey. The length of the survey is projected to be about 12 minutes.
  Intentions to receive COVID-19 vaccines as they are continually recommended will be measured using the Precaution Adoption Process Model (PAPM). The PAPM is a stage-based model of health decision-making, and will be adapted to contain the categories: unengaged, undecided, decided to, and decided not to receive recommended COVID-19 vaccines.
  Participants will provide their stage before and after the intervention has been administered, all within the same survey.

CONTACTS AND LOCATIONS:
Overall Officials: Zeev Rosberger, PhD, Principal Investigator — Lady Davis Institute for Medical Research of the Jewish General Hospital
Locations (1):
- Lady Davis Insitutute for Medical Research, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
The consent form, data collection method, and organizational policy means only aggregated data will be shared with other researchers.

REFERENCES:
- [Background] Zhu P, Tatar O, Griffin-Mathieu G, Perez S, Haward B, Zimet G, Tunis M, Dube E, Rosberger Z. The Efficacy of a Brief, Altruism-Eliciting Video Intervention in Enhancing COVID-19 Vaccination Intentions Among a Population-Based Sample of Younger Adults: Randomized Controlled Trial. JMIR Public Health Surveill. 2022 May 30;8(5):e37328. doi: 10.2196/37328. PMID 35544437
- [Background] Zhu P, Tatar O, Haward B, Steck V, Griffin-Mathieu G, Perez S, Dube E, Zimet G, Rosberger Z. Examining an Altruism-Eliciting Video Intervention to Increase COVID-19 Vaccine Intentions in Younger Adults: A Qualitative Assessment Using the Realistic Evaluation Framework. Vaccines (Basel). 2023 Mar 11;11(3):628. doi: 10.3390/vaccines11030628. PMID 36992212
- [Background] Brewer NT, Chapman GB, Rothman AJ, Leask J, Kempe A. Increasing Vaccination: Putting Psychological Science Into Action. Psychol Sci Public Interest. 2017 Dec;18(3):149-207. doi: 10.1177/1529100618760521. PMID 29611455
- [Background] Yuan S, Chu H. Vaccine for yourself, your community, or your country? Examining audiences' response to distance framing of COVID-19 vaccine messages. Patient Educ Couns. 2022 Feb;105(2):284-289. doi: 10.1016/j.pec.2021.08.019. Epub 2021 Aug 25. PMID 34479746
- [Background] Reifferscheid L, Lee JSW, MacDonald NE, Sadarangani M, Assi A, Lemaire-Paquette S, MacDonald SE. Transition to endemic: acceptance of additional COVID-19 vaccine doses among Canadian adults in a national cross-sectional survey. BMC Public Health. 2022 Sep 14;22(1):1745. doi: 10.1186/s12889-022-14025-8. PMID 36104675

DOCUMENTS (1):
  • Informed Consent Form (2023-02-28): https://cdn.clinicaltrials.gov/large-docs/13/NCT05808413/ICF_000.pdf